CLINICAL TRIAL: NCT01050998
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Efficacy and Safety of CAM-3001 in Subjects With Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of CAM-3001 (Drug) in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: MedImmune Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP219
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Mavrilimumab; CAM-3001
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Mavrilimumab 10 mg (Experimental): Mavrilimumab (CAM-3001) 10 milligram (mg) injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
  Interventions: Biological: Mavrilimumab 10 mg
- Mavrilimumab 30 mg (Experimental): Mavrilimumab (CAM-3001) 30 mg injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
  Interventions: Biological: Mavrilimumab 30 mg
- Mavrilimumab 50 mg (Experimental): Mavrilimumab (CAM-3001) 50 mg injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
  Interventions: Biological: Mavrilimumab 50 mg
- Mavrilimumab 100 mg (Experimental): Mavrilimumab (CAM-3001) 100 mg injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
  Interventions: Biological: Mavrilimumab 100 mg
- Placebo (Placebo Comparator): Placebo matched to mavrilimumab injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mavrilimumab 10 mg — Mavrilimumab (CAM-3001) 10 mg injection subcutaneously every other week for 12 weeks.
  Other Names: CAM-3001
  Arms: Mavrilimumab 10 mg
Biological: Mavrilimumab 30 mg — Mavrilimumab (CAM-3001) 30 mg injection subcutaneously every other week for 12 weeks.
  Other Names: CAM-3001
  Arms: Mavrilimumab 30 mg
Biological: Mavrilimumab 50 mg — Mavrilimumab (CAM-3001) 50 mg injection subcutaneously every other week for 12 weeks.
  Other Names: CAM-3001
  Arms: Mavrilimumab 50 mg
Biological: Mavrilimumab 100 mg — Mavrilimumab (CAM-3001) 100 mg injection subcutaneously every other week for 12 weeks.
  Other Names: CAM-3001
  Arms: Mavrilimumab 100 mg
Other: Placebo — Placebo matched to mavrilimumab injection subcutaneously every other week for 12 weeks.
  Arms: Placebo

SUMMARY:
The primary objectives of this study is to assess the safety, tolerability and efficacy of multiple doses of the mavrilimumab (CAM-3001) administered subcutaneously in subjects with moderately active Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, multiple ascending dose study to evaluate the efficacy and safety of multiple doses of the mavrilimumab (CAM-3001) (10 milligram [mg], 30 mg, 50 mg, and 100 mg) administered subcutaneously in adult subjects with moderately active RA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 80 years (20 to 75 years in Japan)
* Written consent
* Diagnosis of adult onset Rheumatoid Arthritis (RA) of at least 3 months duration as defined by the 1987 American College of Rheumatology (ACR) classification criteria (Arnett et al, 1988)
* Treatment with methotrexate at a stable and tolerated doses
* Positive anti-cyclic citrullinated peptide (CCP) immuno-globulin G antibodies (more than [>] 5 international unit per milliliter [IU/mL]) and/or rheumatoid factor (RF >14 IU/mL) at screening
* Received more than or equal to (>=) 5 milligram (mg) per week folic acid as a single or divided dose during the study.

Exclusion Criteria:

* A rheumatic autoimmune disease other than RA
* A history of, or current, inflammatory joint disease other than RA or other systemic autoimmune disorder
* Subjects at a high risk of infection
* Subjects (male and female) of reproductive potential who are not willing to use contraception from screening through the end date of the trial
* History of methotrexate or any drug-induced lung fibrosis or pneumonitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2011-06-09 (Actual); Study Completion 2012-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Albulescu, Study Director — MedImmune Ltd
Locations (55):
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Czechia (6):
  - Research Site, Bruntál
  - Research Site, Ostrava - Trebovice
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Research Site, Tallinn, Estonia
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Sopron
  - Research Site, Zalaegerszeg
- Japan (17):
  - Research Site, Chiba
  - Research Site, Chiyoda-ku
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Goshogawara-shi
  - Research Site, Hamamatsu
  - Research Site, Iizuka-shi
  - Research Site, Kagoshima
  - Research Site, Kasama-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Nagano
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Omura-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sasebo-shi
  - Research Site, Shinjuku-ku
- Latvia (3):
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Valmiera
- Lithuania (2):
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Legnica
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Torun
  - Research Site, Warsaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Ploieşti
  - Research Site, Târgu Mureş
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Ukraine (3):
  - Research Site, Donetsk
  - Research Site, Kiev
  - Research Site, Kyiv

REFERENCES:
- [Background] Burmester GR, Weinblatt ME, McInnes IB, Porter D, Barbarash O, Vatutin M, Szombati I, Esfandiari E, Sleeman MA, Kane CD, Cavet G, Wang B, Godwood A, Magrini F; EARTH Study Group. Efficacy and safety of mavrilimumab in subjects with rheumatoid arthritis. Ann Rheum Dis. 2013 Sep 1;72(9):1445-52. doi: 10.1136/annrheumdis-2012-202450. Epub 2012 Dec 12. PMID 23234647
- See also: CAM-3001_CP-219_Redacted_4Mar13 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=29&filename=CAM-3001_CP-219_Redacted_4Mar13.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 516 participants were screened out of which 290 participants were randomized in the study.
Period: Overall Study
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg | Placebo
Started | 48 | 49 | 49 | 48 | 96
Completed | 44 | 47 | 46 | 45 | 82
Not Completed | 4 | 2 | 3 | 3 | 14
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 3
Not completed — Other | 3 | 2 | 1 | 1 | 5
Not completed — Data integrity issues | 0 | 0 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population constituted all participants who were randomized into the study regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg | Placebo | Total
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 92 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.9) | 51.1 (12.1) | 52.7 (10.3) | 50.1 (12.1) | 52.1 (12.8) | 51.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 44 | 40 | 82 | 248
  Male | 9 | 6 | 4 | 7 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score of 28 Joints Using C-Reactive Protein (DAS28 [CRP]) Response at Day 85
Description: DAS28 (CRP) calculated swollen joint count (SJC) and tender joint count (TJC) using the 28 joints, general health (GH) using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and CRP (milligram per Liter [mg/L]). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) less than (<) 3.2 = low disease activity, greater than or equal to (>=) 3.2 to 5.1 = moderate to high disease activity and <2.6= remission. A Day 85 responder was defined as a participant who experienced more than 1.2 decrease from baseline in DAS28 (CRP) score at Day 85.
Time Frame: Day 85
Population: The intent-to-treat (ITT) population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants | 32.6 | 37.5 | 63.3 | 47.9 | 68.1
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.578, Fisher Exact; Percent difference = 4.9, 95% CI 2-sided [-11.5 to 22.0] — 95 percent (%) unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p < 0.001, Fisher Exact; Percent difference = 30.7, 95% CI 2-sided [13.4 to 46.3] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.099, Fisher Exact; Percent difference = 15.3, 95% CI 2-sided [-1.6 to 32.2] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p < 0.001, Fisher Exact; Percent difference = 35.5, 95% CI 2-sided [17.8 to 50.6] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001

2. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score of 28 Joints Using C-Reactive Protein (DAS28 [CRP]) Response at Day 85 by Region
Description: DAS28 (CRP) calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and CRP (mg/L). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. A Day 85 responder was defined as a participant who experienced more than 1.2 decrease from baseline in DAS28 (CRP) score at Day 85. DAS28 (CRP) response at Day 85 for the European and Japanese regions were reported.
Time Frame: Day 85
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues. Here "n" signifies participants who were evaluable for the specified region for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  European Region (n=75, 39, 41, 39, 39) | 34.7 | 41.0 | 61.0 | 51.3 | 66.7
  Japanese Region (n=17, 9, 8, 9, 8) | 23.5 | 22.2 | 75.0 | 33.3 | 75.0
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.543, Fisher Exact; Percent difference = 6.4, 95% CI 2-sided [-11.9 to 25.4] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.011, Fisher Exact; Percent difference = 26.3, 95% CI 2-sided [7.2 to 43.6] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.108, Fisher Exact; Percent difference = 16.6, 95% CI 2-sided [-2.5 to 35.5] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.001, Fisher Exact; Percent difference = 32.0, 95% CI 2-sided [12.5 to 49.0] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = -1.3, 95% CI 2-sided [-33.7 to 35.7] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg vs Mavrilimumab 100 mg; Japanese region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.028, Fisher Exact; Percent difference = 51.5, 95% CI 2-sided [8.2 to 77.0] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.661, Fisher Exact; Percent difference = 9.8, 95% CI 2-sided [-24.3 to 46.9] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001

3. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score of 28 Joints Using Erythrocyte Sedimentation Rate (DAS28 [ESR]) at Day 85
Description: DAS28 (ESR) calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]). Total score range: 0-9.4, higher score = more disease activity. DAS28 (ESR) <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. A Day 85 responder was defined as a participant who experienced more than 1.2 decrease from baseline in DAS28 (ESR) score at Day 85.
Time Frame: Day 85
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants | 37.0 | 50.0 | 61.2 | 58.3 | 66.0
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.152, Fisher Exact; Percent difference = 13.0, 95% CI 2-sided [-4.2 to 30.3] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.008, Fisher Exact; Percent difference = 24.3, 95% CI 2-sided [7.0 to 40.3] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.020, Fisher Exact; Percent difference = 21.4, 95% CI 2-sided [3.9 to 37.8] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.002, Fisher Exact; Percent difference = 29.0, 95% CI 2-sided [11.3 to 45.0] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001

4. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score of 28 Joints Using Erythrocyte Sedimentation Rate (DAS28 [ESR]) at Day 85 by Region
Description: DAS28 (ESR) calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]). Total score range: 0-9.4, higher score = more disease activity. DAS28 (ESR) <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. A Day 85 responder was defined as a participant who experienced more than 1.2 decrease from baseline in DAS28 (ESR) score at Day 85. DAS28 (ESR) response at Day 85 for the European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  European Region (n=75, 39, 41, 39, 39) | 41.3 | 51.3 | 58.5 | 61.5 | 64.1
  Japanese Region (n=17, 9, 8, 9, 8) | 17.6 | 44.4 | 75.0 | 44.4 | 75.0
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.328, Fisher Exact; Percent difference = 9.9, 95% CI 2-sided [-9.3 to 29.4] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.084, Fisher Exact; Percent difference = 17.2, 95% CI 2-sided [-2.0 to 35.6] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.049, Fisher Exact; Percent difference = 20.2, 95% CI 2-sided [0.7 to 38.2] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; European region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.030, Fisher Exact; Percent difference = 22.8, 95% CI 2-sided [3.2 to 40.7] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg vs Mavrilimumab 50 mg; Japanese region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.188, Fisher Exact; Percent difference = 26.8, 95% CI 2-sided [-9.3 to 60.7] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg vs Mavrilimumab 100 mg; Japanese region: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.010, Fisher Exact; Percent difference = 57.4, 95% CI 2-sided [15.2 to 81.8] — 95% unconditional exact confidence interval calculated using the method of Agresti and Min, 2001

5. Primary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) Response by European League Against Rheumatism (EULAR) Category at Day 85
Description: DAS28 (CRP) response by EULAR category were used to measure individual response as none, moderate, and good, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with baseline DAS28 (CRP) <3.2; moderate response: change from baseline >1.2 with baseline DAS28 (CRP) >=3.2 to less than or equal to (=<) 5.1 or change from baseline >=0.6 to =< 1.2 with baseline DAS28 (CRP) >=3.2 to =<5.1; no response: change from baseline <0.6 or change from baseline >=0.6 and =<1.2 with baseline DAS28 (CRP) >5.1.
Time Frame: Day 85
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  No response | 51.1 | 47.9 | 28.6 | 35.4 | 23.4
  Moderate response | 34.8 | 31.3 | 38.8 | 41.7 | 42.6
  Good response | 14.1 | 20.8 | 32.7 | 22.9 | 34.0

6. Primary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) Response by European League Against Rheumatism (EULAR) Category at Day 85 by Region
Description: DAS28 (CRP) response by EULAR category were used to measure individual response as none, moderate, and good, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with baseline DAS28 (CRP) <3.2; moderate response: change from baseline >1.2 with baseline DAS28 (CRP) >=3.2 to =< 5.1 or change from baseline >=0.6 to =< 1.2 with baseline DAS28 (CRP) >=3.2 to =<5.1; no response: change from baseline <0.6 or change from baseline >=0.6 and =<1.2 with baseline DAS28 (CRP) >5.1. DAS28 (CRP) response by EULAR category at Day 85 for the European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  European: No response (n=75,39,41,39,39) | 49.3 | 46.2 | 29.3 | 33.3 | 23.1
  European: Moderate response (n=75,39,41,39,39) | 36.0 | 33.3 | 41.5 | 41.0 | 46.2
  European: Good response (n=75,39,41,39,39) | 14.7 | 20.5 | 29.3 | 25.6 | 30.8
  Japanese: No response (n=17,9,8,9,8) | 58.8 | 55.6 | 25.0 | 44.4 | 25.0
  Japanese: Moderate response (n=17,9,8,9,8) | 29.4 | 22.2 | 25.0 | 44.4 | 25.0
  Japanese: Good response (n=17,9,8,9,8) | 11.8 | 22.2 | 50.0 | 11.1 | 50.0

7. Primary Outcome: Percentage of Participants Who Achieved DAS28 (ESR) Response by European League Against Rheumatism (EULAR) Category at Day 85
Description: DAS28 (ESR) response by EULAR category were used to measure individual response as none, moderate, and good, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with baseline DAS28 (ESR) <3.2; moderate response: change from baseline >1.2 with baseline DAS28 (ESR) >=3.2 to =< 5.1 or change from baseline >=0.6 to =< 1.2 with baseline DAS28 (ESR) >=3.2 to =<5.1; no response: change from baseline <0.6 or change from baseline >=0.6 and =<1.2 with baseline DAS28 (ESR) >5.1.
Time Frame: Day 85
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  No response | 55.4 | 39.6 | 36.7 | 33.3 | 25.5
  Moderate response | 35.9 | 45.8 | 44.9 | 54.2 | 53.2
  Good response | 8.7 | 14.6 | 18.4 | 12.5 | 21.3

8. Primary Outcome: Percentage of Participants Who Achieved DAS28 (ESR) Response by European League Against Rheumatism (EULAR) Category at Day 85 by Region
Description: DAS28 (ESR) response by EULAR category were used to measure individual response as none, moderate, and good, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with baseline DAS28 (ESR) <3.2; moderate response: change from baseline >1.2 with baseline DAS28 (ESR) >=3.2 to =< 5.1 or change from baseline >=0.6 to =< 1.2 with baseline DAS28 (ESR) >=3.2 to =<5.1; no response: change from baseline <0.6 or change from baseline >=0.6 and =<1.2 with baseline DAS28 (ESR) >5.1. DAS28 (ESR) response by EULAR category at Day 85 for the European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  European: No response (n=75,39,41,39,39) | 53.3 | 38.5 | 39.0 | 33.3 | 28.2
  European: Moderate response (n=75,39,41,39,39) | 38.7 | 46.2 | 43.9 | 53.8 | 51.3
  European: Good response (n=75,39,41,39,39) | 8.0 | 15.4 | 17.1 | 12.8 | 20.5
  Japanese: No response (n=17,9,8,9,8) | 64.7 | 44.4 | 25.0 | 33.3 | 12.5
  Japanese: Moderate response (n=17,9,8,9,8) | 23.5 | 44.4 | 50.0 | 55.6 | 62.5
  Japanese: Good response (n=17,9,8,9,8) | 11.8 | 11.1 | 25.0 | 11.1 | 25.0

9. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up Day 169 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Day 169 (follow-up)
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
participants
  TEAEs | 46 | 33 | 31 | 26 | 28
  TESAEs | 1 | 2 | 2 | 1 | 0

10. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included blood pressure, pulse rate, temperature, and respiration rate. Vital signs abnormalities reported as TEAEs were reported.
Time Frame: Baseline up to Day 169 (follow-up)
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
participants
  Pyrexia | 1 | 0 | 0 | 2 | 0
  Hypertension | 2 | 0 | 1 | 0 | 0

11. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Results
Description: 12-lead ECG was recorded and corrected QT (QTc) interval was measured with the participant in a rested supine position for at least 10 minutes. Any ECG abnormality deemed clinically significant as per investigator's discretion were reported.
Time Frame: Baseline up to Day 169 (follow-up)
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
participants | 0 | 1 | 0 | 0 | 2

12. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) at Day 85
Description: FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Day 85
Population: The safety population included all participants who received any dose of investigational product. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 87 | 46 | 47 | 49 | 47
liters
  FEV1 | 2.730 (0.764) | 2.877 (0.821) | 2.949 (0.722) | 2.701 (0.489) | 2.793 (0.690)
  FVC | 3.439 (0.949) | 3.582 (0.967) | 3.667 (0.882) | 3.370 (0.527) | 3.499 (0.766)

13. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) at Day 85 by Region
Description: FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FEV1 and FVC at Day 85 for the European and Japanese regions were reported.
Time Frame: Day 85
Population: The safety population included all participants who received any dose of investigational product. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for the specified region for each arm, respectively.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 87 | 46 | 47 | 49 | 47
liters
  European: FEV1 (n=71,37,39,40,39) | 2.811 (0.790) | 2.902 (0.810) | 3.042 (0.745) | 2.698 (0.501) | 2.848 (0.699)
  European: FVC (n=71,37,39,40,39) | 3.537 (0.996) | 3.632 (0.948) | 3.779 (0.917) | 3.355 (0.537) | 3.553 (0.772)
  Japanese: FEV1 (n=16,9,8,9,8) | 2.367 (0.510) | 2.774 (0.908) | 2.493 (0.354) | 2.712 (0.457) | 2.520 (0.616)
  Japanese: FVC (n=16,9,8,9,8) | 3.005 (0.534) | 3.378 (1.076) | 3.119 (0.370) | 3.434 (0.505) | 3.235 (0.725)

14. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) at Day 85
Description: as for outcome 12
Time Frame: Baseline and Day 85
Population: The safety population included all participants who received any dose of investigational product. Here "n" signifies participants who were evaluable for this measure at the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
liters
  Baseline: FEV1 (n=87,43,45,49,48) | 2.790 (0.770) | 2.788 (0.773) | 2.990 (0.765) | 2.760 (0.430) | 2.831 (0.681)
  Change at Day 85: FEV1 (n=87,46,47,49,47) | -0.039 (0.234) | 0.044 (0.231) | 0.016 (0.196) | -0.059 (0.249) | -0.049 (0.221)
  Baseline: FVC (n=87,43,45,49,48) | 3.456 (0.948) | 3.486 (0.963) | 3.759 (0.868) | 3.409 (0.496) | 3.506 (0.804)
  Change at Day 85: FVC (n=87,46,47,49,47) | -0.012 (0.301) | 0.048 (0.243) | -0.013 (0.239) | -0.039 (0.268) | -0.017 (0.218)

15. Primary Outcome: Diffusing Capacity for Carbon Monoxide (DLCO) at Day 85
Description: DLCO is a pulmonary function test that measures the partial pressure difference between inspired and expired carbon monoxide.
Time Frame: Day 85
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent diffusion capacity
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 87 | 46 | 47 | 49 | 47
percent diffusion capacity | 91.7 (16.7) | 95.0 (16.2) | 95.0 (15.1) | 95.0 (15.7) | 89.3 (12.0)

16. Primary Outcome: Diffusing Capacity for Carbon Monoxide (DLCO) at Day 85 by Region
Description: DLCO is a pulmonary function test, and measures the partial pressure difference between inspired and expired carbon monoxide. DLCO% for the European and Japanese regions were reported.
Time Frame: Day 85
Population: The safety population included all participants who received any dose of investigational product. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for this measure for the specified region for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent diffusion capacity
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 87 | 46 | 47 | 49 | 47
percent diffusion capacity
  European region: (n=71,37,39,40,39) | 90.4 (16.5) | 96.0 (16.9) | 94.0 (15.2) | 94.8 (16.5) | 88.6 (10.7)
  Japanese region (n=16,9,8,9,8) | 97.6 (16.9) | 91.0 (13.3) | 100.1 (14.6) | 96.0 (12.6) | 93.0 (17.2)

17. Primary Outcome: Change From Baseline in Diffusing Capacity for Carbon Monoxide (DLCO) at Day 85
Description: DLCO is a pulmonary function test, and measures the partial pressure difference between inspired and expired carbon monoxide.
Time Frame: Baseline and Day 85
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent diffusion capacity
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
percent diffusion capacity
  Baseline (n=86,40,45,49,48) | 91.5 (12.5) | 96.3 (17.7) | 93.7 (15.5) | 97.5 (14.8) | 92.5 (13.7)
  Change at Day 85 (n=87,46,47,49,47) | 0.1 (14.3) | -3.1 (17.3) | 0.4 (11.1) | -2.5 (10.8) | -3.7 (11.3)

18. Primary Outcome: Dyspnea Score at Day 85
Description: Modified Borg dyspnea scale is a validated participant reported outcome assessing participant's perceived difficulty in breathing (dyspnea). The scale ranges from 0 (nothing at all) to 10 (maximal difficulty). Higher scores indicate greater difficulty in breathing.
Time Frame: Day 85
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 89 | 45 | 47 | 49 | 47
units on a scale | 0.25 (0.48) | 0.13 (0.38) | 0.35 (0.70) | 0.15 (0.44) | 0.35 (0.59)

19. Primary Outcome: Change From Baseline in Dyspnea Score at Day 85
Description: as for outcome 18
Time Frame: Baseline and Day 85
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
units on a scale
  Baseline (n=96,48,49,49,48) | 0.29 (0.58) | 0.26 (0.88) | 0.26 (0.59) | 0.19 (0.49) | 0.32 (0.59)
  Change at Day 85 (n=89,45,47,49,47) | -0.06 (0.53) | -0.14 (0.62) | 0.10 (0.44) | -0.04 (0.35) | 0.02 (0.56)

20. Primary Outcome: Categorized Dyspnea Score at Day 85
Description: Modified Borg dyspnea scale is a validated participant reported outcome assessing participant's perceived difficulty in breathing (dyspnea). The scale ranges from 0 (nothing at all) to 10 (maximal difficulty). Higher scores indicate greater difficulty in breathing. The modified BORG dyspnea scale was categorized as - no/slight (0 to 2), moderate (3 and 4), severe (5 and 6) and very severe breathlessness (7 and above).
Time Frame: Day 85
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 89 | 45 | 47 | 49 | 47
participants
  No/Slight breathlessness | 89 (0.58) | 45 (0.88) | 45 (0.59) | 49 (0.49) | 46 (0.59)
  Moderate breathlessness | 0 (0.53) | 0 (0.62) | 2 (0.44) | 0 (0.35) | 1 (0.56)
  Severe breathlessness | 0 | 0 | 0 | 0 | 0
  Very severe breathlessness | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Oxygen Saturation Level at Day 85
Description: Oxygen saturation measured by pulse oximetry which measures the concentration of oxygen in the blood.
Time Frame: Day 85
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 88 | 45 | 47 | 49 | 47
percent saturation | 97.5 (1.2) | 97.6 (1.3) | 97.7 (1.3) | 97.2 (1.8) | 97.3 (1.5)

22. Primary Outcome: Oxygen Saturation Level at Day 85 by Region
Description: Oxygen saturation measured by pulse oximetry which measures the concentration of oxygen in the blood. Oxygen saturation for the European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 88 | 45 | 47 | 49 | 47
percent saturation
  European region: (n=72,36,39,40,39) | 97.5 (1.3) | 97.6 (1.3) | 97.6 (1.3) | 97.2 (2.0) | 97.3 (1.6)
  Japanese region: (n=16,9,8,9,8) | 97.6 (0.9) | 97.4 (1.0) | 98.4 (1.1) | 97.4 (0.7) | 97.3 (1.3)

23. Primary Outcome: Change From Baseline in Oxygen Saturation Level at Day 85
Description: Oxygen saturation measured by pulse oximetry which measures the concentration of oxygen in the blood.
Time Frame: Baseline and Day 85
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
percent saturation
  Baseline (n=96,48,49,49,48) | 97.5 (1.3) | 97.8 (1.6) | 97.6 (1.2) | 97.6 (1.4) | 97.2 (1.7)
  Change at Day 85 (n=88,45,47,49,47) | 0.0 (1.5) | -0.2 (1.5) | 0.1 (1.4) | -0.3 (1.9) | 0.1 (2.1)

24. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Any medically significant change in laboratory evaluations were recorded as adverse events. Following parameters were analyzed for laboratory examination: hematology (haemoglobin, reticulocytes, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes, mean corpuscular volume, mean corpuscular haemoglobin concentration); serum chemistry (creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, gamma glutamyl transferase, CRP, ESR, albumin, total cholesterol, triglycerides, rheumatoid factor and anti-cyclic citrullinated peptide antibodies); urinalysis (albumin, glucose, protein, blood, nitrite).
Time Frame: Baseline up to Day 169 (follow-up)
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
participants
  Blood and lymphatic system disorders | 10 | 3 | 3 | 3 | 4
  Hepatic abnormality | 3 | 5 | 3 | 2 | 3
  Blood cholesterol increased | 0 | 0 | 0 | 1 | 0
  Blood triglycerides increased | 1 | 0 | 0 | 0 | 0
  Hypercholesterolemia | 1 | 1 | 1 | 1 | 0
  Hyperglycemia | 1 | 0 | 0 | 1 | 0
  Urinalysis abnormalities | 3 | 0 | 3 | 1 | 0

25. Secondary Outcome: Change From Baseline in DAS28 (CRP) and DAS28 (ESR) at Day 85
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission.
Time Frame: Baseline and Day 85
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
units on a scale
  DAS28(CRP): Baseline (n=92,48,49,48,47) | 5.43 (0.110) | 5.24 (0.160) | 5.42 (0.139) | 5.14 (0.146) | 5.34 (0.115)
  DAS28(CRP): Change at Day 85 (n=84,45,46,48,46) | -0.97 (0.120) | -1.27 (0.166) | -1.63 (0.163) | -1.32 (0.162) | -1.70 (0.165)
  DAS28(ESR): Baseline: (n=92,48,49,48,47) | 6.18 (0.118) | 6.06 (0.165) | 6.31 (0.145) | 5.98 (0.163) | 6.06 (0.119)
  DAS28(ESR): Change at Day 85 (n=85,45,47,48,46) | -1.04 (0.125) | -1.39 (0.172) | -1.80 (0.170) | -1.46 (0.168) | -1.84 (0.172)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.137, Repeated measures model; Adjusted mean difference = -0.31, 95% CI 2-sided [-0.71 to 0.10], Standard Error of Mean 0.205 — An estimate of the treatment difference and its 95% CI was computed by means of repeated measures model, adjusted for baseline and including a treatment by visit interaction term. Differences <0 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.001, Repeated measures model; Adjusted mean difference = -0.67, 95% CI 2-sided [-1.07 to -0.27], Standard Error of Mean 0.202 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.080, Repeated measures model; Adjusted mean difference = -0.35, 95% CI 2-sided [-0.75 to 0.04], Standard Error of Mean 0.201 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -0.74, 95% CI 2-sided [-1.14 to -0.33], Standard Error of Mean 0.204 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.107, Repeated measures model; Adjusted mean difference = -0.34, 95% CI 2-sided [-0.76 to 0.08], Standard Error of Mean 0.212 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -0.76, 95% CI 2-sided [-1.17 to -0.35], Standard Error of Mean 0.210 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.046, Repeated measures model; Adjusted mean difference = -0.42, 95% CI 2-sided [-0.83 to -0.01], Standard Error of Mean 0.209 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -0.80, 95% CI 2-sided [-1.22 to -0.38], Standard Error of Mean 0.212 — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Change From Baseline in DAS28 (CRP) and DAS28 (ESR) at Day 85 by Region
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. DAS28 (CRP) and DAS28 (ESR) for the European and Japanese regions were reported.
Time Frame: Baseline and Day 85
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues. Here "n" signifies participants who were evaluable for this measure for the specified region for each arm, respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
units on a scale
  European: DAS28(CRP): Baseline (n=75,39,41,39,39) | 5.58 (0.117) | 5.30 (0.172) | 5.48 (0.154) | 5.33 (0.155) | 5.41 (0.111)
  European: DAS28(CRP): Day 85 (n=68,36,38,39,38) | -1.00 (0.133) | -1.40 (0.187) | -1.55 (0.181) | -1.43 (0.181) | -1.70 (0.183)
  Japanese: DAS28(CRP): Baseline (n=17,9,8,9,8) | 4.75 (0.242) | 5.00 (0.427) | 5.12 (0.306) | 4.32 (0.268) | 5.04 (0.413)
  Japanese: DAS28(CRP): Day 85 (n=16,9,8,9,8) | -0.85 (0.281) | -0.73 (0.358) | -2.04 (0.381) | -0.89 (0.361) | -1.71 (0.380)
  European: DAS28(ESR): Baseline (n=75,39,41,39,39) | 6.36 (0.124) | 6.10 (0.180) | 6.36 (0.163) | 6.23 (0.159) | 6.12 (0.118)
  European: DAS28(ESR): Day 85 (n=69,36,39,39,38) | -1.12 (0.140) | -1.51 (0.196) | -1.76 (0.190) | -1.53 (0.190) | -1.85 (0.193)
  Japanese: DAS28(ESR): Baseline (n=17,9,8,9,8) | 5.38 (0.248) | 5.87 (0.426) | 6.05 (0.309) | 4.93 (0.379) | 5.78 (0.404)
  Japanese: DAS28(ESR): Day 85 (n=16,9,8,9,8) | -0.74 (0.276) | -0.83 (0.359) | -1.99 (0.382) | -1.24 (0.362) | -1.78 (0.380)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; European region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.086, Repeated measures model; Adjusted mean difference = -0.40, 95% CI 2-sided [-0.85 to 0.06], Standard Error of Mean 0.230 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; European region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.016, Repeated measures model; Adjusted mean difference = -0.55, 95% CI 2-sided [-0.99 to -0.10], Standard Error of Mean 0.225 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; European region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.059, Repeated measures model; Adjusted mean difference = -0.43, 95% CI 2-sided [-0.87 to 0.02], Standard Error of Mean 0.225 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; European region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.002, Repeated measures model; Adjusted mean difference = -0.70, 95% CI 2-sided [-1.14 to -0.25], Standard Error of Mean 0.227 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; European region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.107, Repeated measures model; Adjusted mean difference = -0.39, 95% CI 2-sided [-0.87 to 0.09], Standard Error of Mean 0.241 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; European region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.007, Repeated measures model; Adjusted mean difference = -0.64, 95% CI 2-sided [-1.11 to -0.18], Standard Error of Mean 0.236 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; European region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.084, Repeated measures model; Adjusted mean difference = -0.41, 95% CI 2-sided [-0.88 to 0.06], Standard Error of Mean 0.236 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; European region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.002, Repeated measures model; Adjusted mean difference = -0.73, 95% CI 2-sided [-1.20 to -0.26], Standard Error of Mean 0.238 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.785, Repeated measures model; Adjusted mean difference = 0.12, 95% CI 2-sided [-0.78 to 1.02], Standard Error of Mean 0.447 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.014, Repeated measures model; Adjusted mean difference = -1.19, 95% CI 2-sided [-2.13 to -0.26], Standard Error of Mean 0.465 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.931, Repeated measures model; Adjusted mean difference = -0.04, 95% CI 2-sided [-0.94 to 0.86], Standard Error of Mean 0.448 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: Analysis reported for change from baseline in DAS28 (CRP) at Day 85; Test type: Superiority or Other; p = 0.070, Repeated measures model; Adjusted mean difference = -0.86, 95% CI 2-sided [-1.80 to 0.07], Standard Error of Mean 0.465 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.854, Repeated measures model; Adjusted mean difference = -0.08, 95% CI 2-sided [-0.99 to 0.82], Standard Error of Mean 0.449 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.011, Repeated measures model; Adjusted mean difference = -1.25, 95% CI 2-sided [-2.19 to -0.31], Standard Error of Mean 0.468 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.271, Repeated measures model; Adjusted mean difference = -0.50, 95% CI 2-sided [-1.40 to 0.40], Standard Error of Mean 0.448 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: Analysis reported for change from baseline in DAS28 (ESR) at Day 85; Test type: Superiority or Other; p = 0.031, Repeated measures model; Adjusted mean difference = -1.03, 95% CI 2-sided [-1.97 to -0.10], Standard Error of Mean 0.465 — [estimate comment as in outcome 25, analysis 1]

27. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) and DAS28 (ESR) Remission at Day 85
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Remission was defined as less than 2.6 DAS28 (ESR) or DAS28 (CRP) score.
Time Frame: Day 85
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  DAS28(CRP) | 7.6 (0.110) | 14.6 (0.160) | 22.4 (0.139) | 18.8 (0.146) | 23.4 (0.115)
  DAS28(ESR) | 3.3 (0.120) | 6.3 (0.166) | 8.2 (0.163) | 8.3 (0.162) | 6.4 (0.165)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; DAS28 (CRP): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.238, Fisher Exact; Percent difference = 7.0, 95% CI 2-sided [-3.3 to 20.5] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; DAS28 (CRP): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.017, Fisher Exact; Percent difference = 14.8, 95% CI 2-sided [2.8 to 29.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; DAS28 (CRP): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.090, Fisher Exact; Percent difference = 11.1, 95% CI 2-sided [0.0 to 25.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; DAS28 (CRP): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.015, Fisher Exact; Percent difference = 15.8, 95% CI 2-sided [2.9 to 31.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; DAS28 (ESR): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.412, Fisher Exact; Percent difference = 3.0, 95% CI 2-sided [-4.2 to 14.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; DAS28 (ESR): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.237, Fisher Exact; Percent difference = 4.9, 95% CI 2-sided [-2.9 to 16.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; DAS28 (ESR): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.231, Fisher Exact; Percent difference = 5.1, 95% CI 2-sided [-2.8 to 16.8] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; DAS28 (ESR): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.406, Fisher Exact; Percent difference = 3.1, 95% CI 2-sided [-4.1 to 14.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001

28. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) and DAS28 (ESR) Remission at Day 85 by Region
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Remission was defined as less than 2.6 DAS28 (ESR) or DAS28 (CRP) score. DAS28 (CRP) and DAS28 (ESR) for the European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  European: DAS28(CRP):(n=75,39,41,39,39) | 6.7 (0.110) | 15.4 (0.160) | 17.1 (0.139) | 17.9 (0.146) | 23.1 (0.115)
  European: DAS28(ESR):(n=75,39,41,39,39) | 1.3 (0.120) | 7.7 (0.166) | 9.8 (0.163) | 7.7 (0.162) | 7.7 (0.165)
  Japanese: DAS28(CRP) (n=17,9,8,9,8) | 11.8 | 11.1 | 50.0 | 22.2 | 25.0
  Japanese: DAS28(ESR) (n=17,9,8,9,8) | 11.8 | 0.0 | 0.0 | 11.1 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; European region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.182, Fisher Exact; Percent difference = 8.7, 95% CI 2-sided [-2.7 to 24.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; European region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.110, Fisher Exact; Percent difference = 10.4, 95% CI 2-sided [-1.2 to 25.5] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; European region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.104, Fisher Exact; Percent difference = 11.3, 95% CI 2-sided [-0.6 to 26.9] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; European region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.016, Fisher Exact; Percent difference = 16.4, 95% CI 2-sided [3.5 to 32.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg vs Mavrilimumab 50 mg vs Mavrilimumab 100 mg; European region (DAS28 [ESR]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.115, Fisher Exact; Percent difference = 6.4, 95% CI 2-sided [-1.0 to 19.3] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; European region (DAS28 [ESR]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.052, Fisher Exact; Percent difference = 8.4, 95% CI 2-sided [0.6 to 21.6] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = -0.7, 95% CI 2-sided [-27.0 to 34.8] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.059, Fisher Exact; Percent difference = 38.2, 95% CI 2-sided [1.6 to 71.2] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 9: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.591, Fisher Exact; Percent difference = 10.5, 95% CI 2-sided [-18.2 to 46.2] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 10: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region (DAS28 [CRP]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.570, Fisher Exact; Percent difference = 13.2, 95% CI 2-sided [-16.6 to 51.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 11: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region (DAS28 [ESR]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.529, Fisher Exact; Percent difference = -11.8, 95% CI 2-sided [-35.0 to 22.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 12: Comparison: Placebo vs Mavrilimumab 30 mg vs Mavrilimumab 100 mg; Japanese region (DAS28 [ESR]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = -11.8, 95% CI 2-sided [-37.5 to 22.6] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 13: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region (DAS28 [ESR]): p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = -0.7, 95% CI 2-sided [-27.0 to 34.8] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001

29. Secondary Outcome: Time to Onset for DAS28 (CRP) and DAS (ESR) Response and Remission
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Response was defined as 1.2 decrease from baseline in DAS28 (CRP) or DAS28 (ESR) score. Remission was defined as less than 2.6 DAS28 (CRP) or DAS28 (ESR) score.
Time Frame: Baseline up to Day 169 (follow-up)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
days
  DAS28 (CRP) Response | 88.0 (0.110) [57.0 to 88.0] | 84.0 (0.160) [43.0 to NA] — Upper limit of CI was not estimable since low number of participants achieved response in this arm. | 43.0 (0.139) [29.0 to 58.0] | 71.0 (0.146) [42.0 to 89.0] | 42.0 (0.115) [29.0 to 45.0]
  DAS28 (CRP) Remission | NA (0.120) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA (0.166) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA (0.163) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA (0.162) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA (0.165) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group.
  DAS28 (ESR) Response | 85.0 [57.0 to 88.0] | 58.0 [43.0 to 86.0] | 30.0 [29.0 to 43.0] | 57.0 [29.0 to 71.0] | 29.0 [28.0 to 42.0]
  DAS28 (ESR) Remission | NA [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group. | NA [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved remission in this group.
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.604, Log Rank; Percent difference
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg vs Mavrilimumab 100 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p < 0.001, Log Rank
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.145, Log Rank
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.282, Log Rank
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 30 mg vs Mavrilimumab 100 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p < 0.001, Log Rank
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.047, Log Rank

30. Secondary Outcome: Time to Onset for DAS28 (CRP) and DAS (ESR) Response and Remission by Region
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Response was defined as 1.2 decrease from baseline in DAS28 (CRP) or DAS28 (ESR) score. Remission was defined as less than 2.6 DAS28 (CRP) or DAS28 (ESR) score. Time to response for DAS28 (CRP) and DAS28 (ESR) by region were reported. Time to remission for DAS28 (CRP) and DAS28 (ESR) by region were not analyzed because time to remission for the overall study population could not be achieved.
Time Frame: Baseline up to Day 169 (follow-up)
Population: as for outcome 26
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
days
  European: DAS28 (CRP) Response (n=75,39,41,39,39) | 85.0 (0.110) [57.0 to 88.0] | 43.0 (0.160) [43.0 to NA] — Upper limit of CI was not estimable since low number of participants achieved response in this arm. | 43.0 (0.139) [42.0 to 71.0] | 50.0 (0.146) [29.0 to 89.0] | 42.0 (0.115) [29.0 to 57.0]
  Japanese: DAS28 (CRP) Response (n=17,9,8,9,8) | NA (0.120) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved response in this group. | NA (0.166) [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved response in this group. | 22.5 (0.163) [15.0 to 57.0] | 87.0 (0.162) [30.0 to 87.0] | 37.0 (0.165) [15.0 to 57.0]
  European: DAS28 (ESR) Response (n=75,39,41,39,39) | 71.0 [57.0 to 88.0] | 57.0 [30.0 to 85.0] | 42.0 [29.0 to 43.0] | 52.5 [29.0 to 84.0] | 29.0 [28.0 to 42.0]
  Japanese: DAS28 (ESR) Response (n=17,9,8,9,8) | NA [NA to NA] — Median and 95% CI were not estimable since less than 50% of the participants achieved response in this group. | 86.0 [57.0 to 86.0] | 29.0 [15.0 to 44.0] | 44.5 [29.0 to NA] — Upper limit of CI was not estimable since low number of participants achieved response in this arm. | 30.0 [15.0 to 44.0]
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; European region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.237, Log Rank; Percent difference
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; European region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.005, Log Rank
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; European region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.134, Log Rank
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; European region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p < 0.001, Log Rank
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.265, Log Rank
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.013, Log Rank
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.952, Log Rank
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.004, Log Rank
Statistical Analysis 9: Comparison: Placebo vs Mavrilimumab 10 mg; European region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.246, Log Rank
Statistical Analysis 10: Comparison: Placebo vs Mavrilimumab 30 mg vs Mavrilimumab 100 mg; European region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p < 0.001, Log Rank
Statistical Analysis 11: Comparison: Placebo vs Mavrilimumab 50 mg; European region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.126, Log Rank
Statistical Analysis 12: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.831, Log Rank
Statistical Analysis 13: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.005, Log Rank
Statistical Analysis 14: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.125, Log Rank
Statistical Analysis 15: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p < 0.001, Log Rank

31. Secondary Outcome: Duration of DAS28 (CRP) and DAS28 (ESR) Response and Remission
Description: DAS28 calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst) and CRP (mg/L) for DAS28 (CRP) or ESR (mm/hour) for DAS28 (ESR). Total score range: 0-9.4, higher score = more disease activity. DAS28 <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Response was defined as 1.2 decrease from baseline in DAS28 (CRP) or DAS28 (ESR) score. Remission was defined as less than 2.6 DAS28 (CRP) or DAS28 (ESR) score. Expected duration of response (DOR) was calculated as response rate (in percentage) multiplied by mean DOR (in days) by using Weibull Model. Duration of DAS28 (CRP) and DAS28 (ESR) remission were not analyzed because very few participants achieved remission in the overall study population.
Time Frame: Baseline up to Day 169
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues. Here "n" signifies participants who were evaluable for this measure for the specified parameter for each arm, respectively.
Measure: Number; unit: Percentage of days
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
Percentage of days
  DAS28 (CRP) Response | 43.40 (0.110) [0.61 to 1.55] | 42.19 (0.160) [43.0 to NA] | 81.89 (0.139) [29.0 to 58.0] | 54.80 (0.146) [42.0 to 89.0] | 83.07 (0.115) [29.0 to 45.0]
  DAS28 (ESR) Response | 46.11 (0.120) [NA to NA] | 52.96 (0.166) [NA to NA] | 71.14 (0.163) [NA to NA] | 75.97 (0.162) [NA to NA] | 96.52 (0.165) [NA to NA]
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.486, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 1.15, 95% CI 2-sided [0.78 to 1.69] — Ratio greater than (>) 1 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.015, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 1.54, 95% CI 2-sided [1.09 to 2.18] — Ratio >1 favored mavrilimumab
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p = 0.006, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 1.65, 95% CI 2-sided [1.15 to 2.36] — Ratio >1 favored mavrilimumab
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for DAS28 (ESR) response; Test type: Superiority or Other; p < 0.001, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 2.09, 95% CI 2-sided [1.49 to 2.93] — Ratio >1 favored mavrilimumab
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.906, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 0.97, 95% CI 2-sided [0.61 to 1.55] — Ratio >1 favored mavrilimumab
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p < 0.001, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 1.89, 95% CI 2-sided [1.31 to 2.71] — Ratio >1 favored mavrilimumab
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p = 0.272, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 1.26, 95% CI 2-sided [0.83 to 1.91] — Ratio >1 favored mavrilimumab
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for DAS28 (CRP) response; Test type: Superiority or Other; p < 0.001, Exponential,Weibull and Log normal model; Ratio of expected duration of response = 1.91, 95% CI 2-sided [1.34 to 2.72] — Ratio >1 favored mavrilimumab

32. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20), ACR50 and ACR70 Responses at Day 85
Description: ACR20, ACR50, and ACR70, were defined as greater than or equal to (>=) 20 percent (%),>=50%, or >=70% improvement, respectively, in: swollen joint count and tender joint count and >=20%, >=50%, or >=70% improvement, respectively, in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Day 85
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  ACR20 | 37.0 (0.110) [57.0 to 88.0] | 41.7 (0.160) [43.0 to NA] | 57.1 (0.139) [29.0 to 58.0] | 37.5 (0.146) [42.0 to 89.0] | 70.2 (0.115) [29.0 to 45.0]
  ACR50 | 12.0 (0.120) [NA to NA] | 20.8 (0.166) [NA to NA] | 30.6 (0.163) [NA to NA] | 16.7 (0.162) [NA to NA] | 34.0 (0.165) [NA to NA]
  ACR70 | 5.4 [57.0 to 88.0] | 4.2 [43.0 to 86.0] | 10.2 [29.0 to 43.0] | 6.3 [29.0 to 71.0] | 14.9 [28.0 to 42.0]
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; ACR20: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.589, Fisher Exact; Percent difference = 4.7, 95% CI 2-sided [-12.1 to 22.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; ACR20: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.032, Fisher Exact; Percent difference = 20.2, 95% CI [2.8 to 36.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; ACR20: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = 0.5, 95% CI 2-sided [-16.0 to 18.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; ACR20: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p < 0.001, Fisher Exact; Percent difference = 33.3, 95% CI 2-sided [15.6 to 48.6] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; ACR50: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.212, Fisher Exact; Percent difference = 8.9, 95% CI 2-sided [-3.5 to 23.6] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; ACR50: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.011, Fisher Exact; Percent difference = 18.7, 95% CI 2-sided [4.8 to 34.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; ACR50: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.446, Fisher Exact; Percent difference = 4.7, 95% CI 2-sided [-7.0 to 19.1] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; ACR50: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.003, Fisher Exact; Percent difference = 22.1, 95% CI 2-sided [7.6 to 37.8] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 9: Comparison: Placebo vs Mavrilimumab 10 mg; ACR70: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = -1.3, 95% CI 2-sided [-8.9 to 9.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 10: Comparison: Placebo vs Mavrilimumab 30 mg; ACR70: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.317, Fisher Exact; Percent difference = 4.8, 95% CI 2-sided [-4.1 to 17.5] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 11: Comparison: Placebo vs Mavrilimumab 50 mg; ACR70: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = 0.8, 95% CI 2-sided [-7.2 to 12.1] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 12: Comparison: Placebo vs Mavrilimumab 100 mg; ACR70: p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.106, Fisher Exact; Percent difference = 9.5, 95% CI 2-sided [-0.5 to 23.5] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001

33. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20), ACR50 and ACR70 Responses at Day 85 by Region
Description: ACR20, ACR50, and ACR70, were defined as >=20%, >=50%, or >=70% improvement, respectively, in: SJC and TJC and >=20%, >=50%, or >=70% improvement, respectively, in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP. Data for the European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
percentage of participants
  European: ACR20 (n=75,39,41,39,39) | 40.0 (0.110) [57.0 to 88.0] | 41.0 (0.160) [43.0 to NA] | 56.1 (0.139) [29.0 to 58.0] | 41.0 (0.146) [42.0 to 89.0] | 69.2 (0.115) [29.0 to 45.0]
  Japanese: ACR20 (n=17,9,8,9,8) | 23.5 (0.120) [NA to NA] | 44.4 (0.166) [NA to NA] | 62.5 (0.163) [NA to NA] | 22.2 (0.162) [NA to NA] | 75.0 (0.165) [NA to NA]
  European: ACR50 (n=75,39,41,39,39) | 12.0 [57.0 to 88.0] | 23.1 [43.0 to 86.0] | 29.3 [29.0 to 43.0] | 20.5 [29.0 to 71.0] | 30.8 [28.0 to 42.0]
  Japanese: ACR50 (n=17,9,8,9,8) | 11.8 [NA to NA] | 11.1 [NA to NA] | 37.5 [NA to NA] | 0.0 [NA to NA] | 50.0 [NA to NA]
  European: ACR70 (n=75,39,41,39,39) | 4.0 | 5.1 | 9.8 | 7.7 | 17.9
  Japanese: ACR70 (n=17,9,8,9,8) | 11.8 | 0.0 | 12.5 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; European region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = 1.0, 95% CI 2-sided [-17.7 to 20.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; European region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.120, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 16.1, 95% CI 2-sided [-3.1 to 34.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; European region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 1.0, 95% CI 2-sided [-17.7 to 20.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; European region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.005, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 29.2, 95% CI 2-sided [9.7 to 46.1] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.382, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 20.9, 95% CI 2-sided [-16.4 to 55.9] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.087, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 39.0, 95% CI 2-sided [-2.7 to 69.6] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = -1.3, 95% CI 2-sided [-33.7 to 35.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: ACR20 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.028, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 51.5, 95% CI 2-sided [8.2 to 77.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 9: Comparison: Placebo vs Mavrilimumab 10 mg; European region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.175, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 11.1, 95% CI 2-sided [-2.9 to 27.9] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 10: Comparison: Placebo vs Mavrilimumab 30 mg; European region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.026, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 17.3, 95% CI 2-sided [2.4 to 34.1] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 11: Comparison: Placebo vs Mavrilimumab 50 mg; European region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.271, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 8.5, 95% CI 2-sided [-5.1 to 24.9] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 12: Comparison: Placebo vs Mavrilimumab 100 mg; European region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.021, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 18.8, 95% CI 2-sided [3.4 to 36.0] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 13: Comparison: Placebo vs Mavrilimumab 10 mg; Japanese region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = -0.7, 95% CI 2-sided [-27.0 to 34.8] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 14: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.283, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 25.7, 95% CI 2-sided [-8.8 to 63.2] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 15: Comparison: Placebo vs Mavrilimumab 50 mg; Japanese region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.529, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = -11.8, 95% CI 2-sided [-35.0 to 22.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 16: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: ACR50 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.059, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 38.2, 95% CI 2-sided [1.6 to 71.2] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 17: Comparison: Placebo vs Mavrilimumab 10 mg; European region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 1.1, 95% CI 2-sided [-7.0 to 14.2] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 18: Comparison: Placebo vs Mavrilimumab 30 mg; European region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.242, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 5.8, 95% CI 2-sided [-3.7 to 19.4] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 19: Comparison: Placebo vs Mavrilimumab 50 mg; European region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.410, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 3.7, 95% CI 2-sided [-5.1 to 16.9] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 20: Comparison: Placebo vs Mavrilimumab 100 mg; European region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.030, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 13.9, 95% CI 2-sided [2.7 to 29.5] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 21: Comparison: Placebo vs Mavrilimumab 10 mg vs Mavrilimumab 50 mg; Japanese region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 0.529, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = -11.8, 95% CI 2-sided [-35.0 to 22.7] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 22: Comparison: Placebo vs Mavrilimumab 30 mg; Japanese region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = 0.7, 95% CI 2-sided [-26.7 to 39.5] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001
Statistical Analysis 23: Comparison: Placebo vs Mavrilimumab 100 mg; Japanese region: ACR70 - p-value was calculated using a two-tailed Fisher's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact; p-value was calculated using a two-tailed Fisher's exact test; Percent difference = -11.8, 95% CI 2-sided [-37.5 to 22.6] — 95% unconditional exact CI was calculated using the method of Agresti and Min, 2001

34. Secondary Outcome: Number of Participants Who Achieved ACR Categorical Responses
Description: ACR20, ACR50, and ACR70, were defined as >=20%, >=50%, or >=70% improvement, respectively, in: SJC and TJC and >=20%, >=50%, or >=70% improvement, respectively, in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP. ACR responses were categorized as "No response", "ACR20 but not ACR50", "ACR50 but not ACR70", and "ACR70".
Time Frame: Day 85
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
participants
  No response | 58 (0.110) [57.0 to 88.0] | 28 (0.160) [43.0 to NA] | 21 (0.139) [29.0 to 58.0] | 30 (0.146) [42.0 to 89.0] | 14 (0.115) [29.0 to 45.0]
  ACR20 but not ACR50 | 23 (0.120) [NA to NA] | 10 (0.166) [NA to NA] | 13 (0.163) [NA to NA] | 10 (0.162) [NA to NA] | 17 (0.165) [NA to NA]
  ACR50 but not ACR70 | 6 [57.0 to 88.0] | 8 [43.0 to 86.0] | 10 [29.0 to 43.0] | 5 [29.0 to 71.0] | 9 [28.0 to 42.0]
  ACR70 | 5 [NA to NA] | 2 [NA to NA] | 5 [NA to NA] | 3 [NA to NA] | 7 [NA to NA]

35. Secondary Outcome: Continuous ACR (ACRn) Score
Description: ACR score - continuous (ACRn) was defined as the minimum of the percentage improvement in TJC, SJC and the median of the percentage improvements in the other five components of the ACR criteria (participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; disability index of the HAQ; and CRP). Total score range was -100 to 100, where negative numbers indicated worsening and positive numbers indicated improvement.
Time Frame: Day 85
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 84 | 44 | 47 | 45 | 46
units on a scale | 5.09 (4.230) [57.0 to 88.0] | 19.13 (5.818) [43.0 to NA] | 26.31 (5.652) [29.0 to 58.0] | 12.17 (5.786) [42.0 to 89.0] | 37.11 (5.723) [29.0 to 45.0]
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; Test type: Superiority or Other; p = 0.051, Repeated measures model; Adjusted Mean difference = 14.05, 95% CI 2-sided [-0.05 to 28.15], Standard Error of Mean 7.162 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.003, Repeated measures model; Adjusted Mean difference = 21.23, 95% CI 2-sided [7.39 to 35.07], Standard Error of Mean 7.028 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; Test type: Superiority or Other; p = 0.322, Repeated measures model; Adjusted Mean difference = 7.09, 95% CI 2-sided [-6.96 to 21.14], Standard Error of Mean 7.136 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted Mean difference = 32.03, 95% CI 2-sided [18.08 to 45.98], Standard Error of Mean 7.085 — [estimate comment as in outcome 25, analysis 1]

36. Secondary Outcome: Continuous ACR (ACRn) Score by Region
Description: ACR score - continuous (ACRn) was defined as the minimum of the percentage improvement in TJC, SJC and the median of the percentage improvements in the other five components of the ACR criteria (participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; disability index of the HAQ; and CRP). Total score range was -100 to 100, where negative numbers indicated worsening and positive numbers indicated improvement. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: ITT population. Six participants were excluded from the ITT population for data integrity issues. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for this measure for the specified region for each arm, respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 84 | 44 | 47 | 45 | 46
units on a scale
  European region (n=69,36,39,38,38) | 4.71 (4.689) [57.0 to 88.0] | 19.18 (6.489) [43.0 to NA] | 24.12 (6.263) [29.0 to 58.0] | 12.53 (6.356) [42.0 to 89.0] | 36.06 (6.356) [29.0 to 45.0]
  Japanese region (n=15,8,8,7,8) | 5.99 (10.060) [NA to NA] | 18.09 (13.843) [NA to NA] | 37.22 (13.843) [NA to NA] | 10.20 (14.799) [NA to NA] | 42.09 (13.843) [NA to NA]
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for European region; Test type: Superiority or Other; p = 0.071, Repeated measures model; Adjusted Mean difference = 14.49, 95% CI 2-sided [-1.24 to 30.22], Standard Error of Mean 7.981 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for European region; Test type: Superiority or Other; p = 0.013, Repeated measures model; Adjusted mean difference = 19.43, 95% CI 2-sided [4.06 to 34.80], Standard Error of Mean 7.798 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for European region; Test type: Superiority or Other; p = 0.320, Repeated measures model; Adjusted mean difference = 7.84, 95% CI 2-sided [-7.68 to 23.36], Standard Error of Mean 7.873 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for European region; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = 31.37, 95% CI 2-sided [15.85 to 46.89], Standard Error of Mean 7.873 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 10 mg; Analysis reported for Japanese region; Test type: Superiority or Other; p = 0.483, Repeated measures model; Adjusted mean difference = 12.11, 95% CI 2-sided [-22.41 to 46.64], Standard Error of Mean 17.089 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for Japanese region; Test type: Superiority or Other; p = 0.075, Repeated measures model; Adjusted mean difference = 31.24, 95% CI 2-sided [-3.28 to 65.77], Standard Error of Mean 17.089 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Mavrilimumab 50 mg; Analysis reported for Japanese region; Test type: Superiority or Other; p = 0.815, Repeated measures model; Adjusted mean difference = 4.22, 95% CI 2-sided [-31.89 to 40.32], Standard Error of Mean 17.872 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for Japanese region; Test type: Superiority or Other; p = 0.041, Repeated measures model; Adjusted mean difference = 36.11, 95% CI 2-sided [1.58 to 70.63], Standard Error of Mean 17.089 — [estimate comment as in outcome 25, analysis 1]

37. Secondary Outcome: Swollen and Tender Joint Count
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1. Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
joints
  Swollen joint count | 9.2 (10.0) [57.0 to 88.0] | 8.0 (8.4) [43.0 to NA] | 5.4 (6.8) [29.0 to 58.0] | 5.8 (7.4) [42.0 to 89.0] | 4.4 (4.3) [29.0 to 45.0]
  Tender joint count | 14.8 (13.1) [NA to NA] | 11.2 (10.9) [NA to NA] | 9.8 (10.1) [NA to NA] | 13.9 (11.8) [NA to NA] | 9.1 (8.8) [NA to NA]

38. Secondary Outcome: Swollen and Tender Joint Count by Region
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1. Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1. Data for the European and Japanese regions were reported.
Time Frame: Day 85
Population: ITT population. Six participants were excluded from the ITT population for data integrity issues. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for the specified region for each arm, respectively.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
joints
  European: Swollen joint count (n=69,36,39,39,38) | 9.6 (10.4) [57.0 to 88.0] | 8.0 (8.2) [43.0 to NA] | 5.6 (7.2) [29.0 to 58.0] | 6.4 (8.0) [42.0 to 89.0] | 4.2 (4.4) [29.0 to 45.0]
  Japanese: Swollen joint count (n=16,9,8,9,8) | 7.6 (8.0) [NA to NA] | 7.8 (9.5) [NA to NA] | 4.6 (4.1) [NA to NA] | 3.1 (2.9) [NA to NA] | 4.9 (4.3) [NA to NA]
  European: Tender joint count (n=69,36,39,39,38) | 15.9 (13.1) [57.0 to 88.0] | 11.0 (11.4) [43.0 to 86.0] | 11.2 (10.5) [29.0 to 43.0] | 14.8 (12.0) [29.0 to 71.0] | 9.9 (9.0) [28.0 to 42.0]
  Japanese: Tender joint count (n=16,9,8,9,8) | 9.6 (11.9) [NA to NA] | 12.1 (9.1) [NA to NA] | 2.8 (2.4) [NA to NA] | 9.6 (10.1) [NA to NA] | 5.5 (7.2) [NA to NA]

39. Secondary Outcome: Physician Global Assessment of Disease Activity Score
Description: Physician Global Assessment of Arthritis was measured on a 0 to 10 centimeter (cm) Visual Analogue Scale (VAS), where 0 cm = very good and 10 cm = very bad.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
cm | 3.82 (2.05) [57.0 to 88.0] | 3.30 (2.16) [43.0 to NA] | 3.13 (1.80) [29.0 to 58.0] | 3.45 (1.97) [42.0 to 89.0] | 2.95 (1.70) [29.0 to 45.0]

40. Secondary Outcome: Physician Global Assessment of Disease Activity Score by Region
Description: Physician Global Assessment of Arthritis was measured on a 0 to 10 cm VAS, where 0 cm = very good and 10 cm = very bad. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
cm
  European region (n=69,36,39,39,38) | 3.93 (2.06) [57.0 to 88.0] | 3.29 (2.21) [43.0 to NA] | 3.20 (1.79) [29.0 to 58.0] | 3.54 (1.98) [42.0 to 89.0] | 3.12 (1.74) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 3.31 (1.99) [NA to NA] | 3.37 (2.05) [NA to NA] | 2.79 (1.91) [NA to NA] | 3.08 (2.03) [NA to NA] | 2.18 (1.37) [NA to NA]

41. Secondary Outcome: Patient Global Assessment of Disease Activity Score
Description: Participants responded to a question, "Considering all the ways your arthritis affects you, how are you feeling today?" by using a 0 - 100 millimeter (mm) VAS, where 0 = very well and 100 = very poorly.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
mm | 45.1 (24.2) [57.0 to 88.0] | 40.0 (22.8) [43.0 to NA] | 37.2 (21.1) [29.0 to 58.0] | 41.1 (23.2) [42.0 to 89.0] | 35.5 (19.3) [29.0 to 45.0]

42. Secondary Outcome: Patient Global Assessment of Disease Activity Score by Region
Description: Participants responded to a question, "Considering all the ways your arthritis affects you, how are you feeling today?" by using a 0 - 100 mm VAS, where 0 = very well and 100 = very poorly. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
mm
  European region (n=69,36,39,39,38) | 45.9 (23.8) [57.0 to 88.0] | 39.5 (22.2) [43.0 to NA] | 39.0 (20.6) [29.0 to 58.0] | 42.5 (23.6) [42.0 to 89.0] | 37.3 (19.2) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 41.5 (26.2) [NA to NA] | 41.9 (26.5) [NA to NA] | 28.8 (22.7) [NA to NA] | 35.0 (21.4) [NA to NA] | 26.9 (18.7) [NA to NA]

43. Secondary Outcome: Patient Pain Assessment Score
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
mm | 44.5 (24.9) [57.0 to 88.0] | 38.7 (24.1) [43.0 to NA] | 38.1 (24.2) [29.0 to 58.0] | 40.1 (24.2) [42.0 to 89.0] | 34.4 (21.6) [29.0 to 45.0]

44. Secondary Outcome: Patient Pain Assessment Score by Region
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
mm
  European region (n=69,36,39,39,38) | 44.9 (24.4) [57.0 to 88.0] | 38.1 (24.1) [43.0 to NA] | 39.1 (24.0) [29.0 to 58.0] | 41.4 (24.4) [42.0 to 89.0] | 36.0 (22.0) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 42.6 (27.8) [NA to NA] | 41.1 (25.5) [NA to NA] | 33.3 (26.1) [NA to NA] | 34.1 (23.6) [NA to NA] | 27.0 (19.4) [NA to NA]

45. Secondary Outcome: Health Assessments Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
units on a scale | 1.19 (0.68) [57.0 to 88.0] | 1.02 (0.51) [43.0 to NA] | 1.02 (0.64) [29.0 to 58.0] | 1.10 (0.61) [42.0 to 89.0] | 0.95 (0.59) [29.0 to 45.0]

46. Secondary Outcome: Health Assessments Questionnaire-Disability Index (HAQ-DI) Score by Region
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
units on a scale
  European region (n=69,36,39,39,38) | 1.22 (0.65) [57.0 to 88.0] | 1.10 (0.47) [43.0 to NA] | 1.05 (0.67) [29.0 to 58.0] | 1.16 (0.63) [42.0 to 89.0] | 1.03 (0.56) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 1.09 (0.82) [NA to NA] | 0.72 (0.61) [NA to NA] | 0.91 (0.53) [NA to NA] | 0.82 (0.44) [NA to NA] | 0.56 (0.60) [NA to NA]

47. Secondary Outcome: Health Assessments Questionnaire (HAQ) Pain Score
Description: Participants were asked to assess the severity of pain in the past week on a 100 VAS with 0 being no pain and 100 being severe pain.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
units on a scale | 46.3 (24.3) [57.0 to 88.0] | 40.9 (23.5) [43.0 to NA] | 39.0 (25.0) [29.0 to 58.0] | 42.6 (23.5) [42.0 to 89.0] | 35.0 (20.8) [29.0 to 45.0]

48. Secondary Outcome: Health Assessments Questionnaire (HAQ) Pain Score by Region
Description: Participants were asked to assess the severity of pain in the past week on a 100 VAS with 0 being no pain and 100 being severe pain. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
units on a scale
  European region (n=69,36,39,39,38) | 47.0 (23.9) [57.0 to 88.0] | 40.3 (23.6) [43.0 to NA] | 40.6 (24.8) [29.0 to 58.0] | 43.8 (23.8) [42.0 to 89.0] | 36.5 (21.1) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 43.1 (26.3) [NA to NA] | 43.1 (24.5) [NA to NA] | 31.0 (26.1) [NA to NA] | 37.3 (22.9) [NA to NA] | 28.3 (19.1) [NA to NA]

49. Secondary Outcome: Serum Concentration of C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 46 | 48 | 46
mg/L | 11.49 (4.67) [57.0 to 88.0] | 9.62 (4.15) [43.0 to NA] | 9.35 (3.92) [29.0 to 58.0] | 5.71 (2.97) [42.0 to 89.0] | 6.12 (2.90) [29.0 to 45.0]

50. Secondary Outcome: Serum Concentration of C-Reactive Protein (CRP) by Region
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 46 | 48 | 46
mg/L
  European region (n=69,36,38,39,38) | 11.89 (18.57) [57.0 to 88.0] | 8.86 (13.10) [43.0 to NA] | 10.24 (16.68) [29.0 to 58.0] | 6.50 (7.60) [42.0 to 89.0] | 5.84 (9.68) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 9.75 (11.93) [NA to NA] | 12.67 (18.47) [NA to NA] | 5.13 (6.83) [NA to NA] | 2.28 (1.92) [NA to NA] | 7.44 (12.26) [NA to NA]

51. Secondary Outcome: Serum Concentration of Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube.
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
mm/hr | 34.4 (26.5) [57.0 to 88.0] | 31.3 (19.0) [43.0 to NA] | 34.1 (23.6) [29.0 to 58.0] | 29.7 (19.1) [42.0 to 89.0] | 23.6 (14.6) [29.0 to 45.0]

52. Secondary Outcome: Serum Concentration of Erythrocyte Sedimentation Rate (ESR) by Region
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Data for European and Japanese regions were reported.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 47 | 48 | 46
mm/hr
  European region (n=69,36,39,39,38) | 33.9 (27.8) [57.0 to 88.0] | 30.3 (18.3) [43.0 to NA] | 33.2 (23.9) [29.0 to 58.0] | 32.7 (19.0) [42.0 to 89.0] | 23.1 (14.3) [29.0 to 45.0]
  Japanese region (n=16,9,8,9,8) | 36.6 (20.8) [NA to NA] | 35.0 (22.5) [NA to NA] | 38.8 (22.6) [NA to NA] | 16.3 (13.6) [NA to NA] | 25.9 (16.7) [NA to NA]

53. Secondary Outcome: Serum Concentration of Rheumatoid Factor (RF)
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units per milliliter
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 85 | 45 | 46 | 48 | 46
units per milliliter | 109.82 (135.39) [57.0 to 88.0] | 79.62 (93.21) [43.0 to NA] | 177.84 (352.16) [29.0 to 58.0] | 85.15 (81.47) [42.0 to 89.0] | 83.26 (118.14) [29.0 to 45.0]

54. Secondary Outcome: Serum Concentration of Anti-Citrullinated-Peptide-Antibody (ACPA)
Time Frame: Day 85
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units per milliliter
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 84 | 45 | 46 | 48 | 45
units per milliliter | 295.90 (920.92) [57.0 to 88.0] | 232.22 (469.86) [43.0 to NA] | 211.77 (250.50) [29.0 to 58.0] | 330.82 (549.05) [42.0 to 89.0] | 221.18 (333.28) [29.0 to 45.0]

55. Secondary Outcome: Number of Participants Who Had Additional Medications
Description: Additional medication included concomitant medication (medication used for purposes other than managing rheumatoid arthritis [RA]) and RA medication (for managing RA). Number of participants who used concomitant medication and RA medication was reported by anatomical therapeutic chemical (ATC) classification system.
Time Frame: Baseline up to Day 169
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
participants
  Concomitant: Blood and blood forming agents | 88 (0.110) [57.0 to 88.0] | 47 (0.160) [43.0 to NA] | 49 (0.139) [29.0 to 58.0] | 47 (0.146) [42.0 to 89.0] | 45 (0.115) [29.0 to 45.0]
  Concomitant: Alimentary tract and metabolism | 45 (0.120) [NA to NA] | 25 (0.166) [NA to NA] | 25 (0.163) [NA to NA] | 28 (0.162) [NA to NA] | 23 (0.165) [NA to NA]
  Concomitant: Cardiovascular system | 30 [57.0 to 88.0] | 20 [43.0 to 86.0] | 19 [29.0 to 43.0] | 12 [29.0 to 71.0] | 22 [28.0 to 42.0]
  Concomitant: Nervous system | 14 [NA to NA] | 9 [NA to NA] | 9 [NA to NA] | 6 [NA to NA] | 3 [NA to NA]
  Concomitant: Musculo-skeletal system | 11 | 9 | 5 | 8 | 5
  Concomitant: Respiratory system | 11 | 6 | 7 | 5 | 5
  Concomitant: Anti-infective for systemic use | 10 | 6 | 6 | 8 | 2
  Concomitant:Genito-urinary system and sex hormones | 4 | 6 | 6 | 4 | 4
  Concomitant: Systemic hormonal preps | 8 | 5 | 4 | 2 | 0
  Concomitant: Various | 6 | 5 | 2 | 2 | 4
  Concomitant: Dermatologicals | 2 | 1 | 5 | 2 | 2
  Concomitant: Sensory organs | 0 | 2 | 3 | 2 | 2
  Concomitant: Anti-parasitic products | 1 | 0 | 0 | 0 | 0
  RA: Antineoplastic and immunomodulating agents | 92 | 48 | 49 | 48 | 47
  RA: Musculo-skeletal system | 65 | 35 | 38 | 32 | 31
  RA: Systemic hormonal preps | 47 | 23 | 21 | 21 | 23
  RA: Nervous system | 4 | 0 | 2 | 2 | 1
  RA: Alimentary tract and metabolism | 0 | 2 | 0 | 1 | 0
  RA: Dermatologicals | 1 | 0 | 0 | 0 | 1
  RA: Respiratory system | 0 | 0 | 0 | 0 | 1
  RA: Sensory organs | 0 | 0 | 0 | 0 | 1

56. Secondary Outcome: Number of Participants With Change in Methotrexate (MTX) and Corticosteroid (CST) Dose
Description: Participants received MTX at stable and tolerated dose during baseline were categorized as "low dose (<12.5 mg per week [mg/wk])", "medium dose (>=12.5 - <20 mg/wk)", and "high dose (>=20 mg/wk)". Participants received oral CST at stable dose during baseline were categorized as "low dose (<5 mg/day)", and "high dose (>=5 mg/day)". Change in MTX and CST dose from baseline between Day 1-85 and Day 86-169 were categorized as follows: 'Increased', 'no change' and 'decreased'. Participants were counted once with dose increases counted first, followed by no change and then dose decreases.
Time Frame: Baseline, Day 1 to 85, Day 86 to 169
Population: The ITT population analysis set included all randomized participants regardless of whether participants received any investigational product. Six participants were excluded from the ITT population for data integrity issues. Here "n" signifies participants who were evaluable for the specified parameter for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 92 | 48 | 49 | 48 | 47
participants
  MTX: Low dose (Baseline) (n=92,48,49,48,47) | 39 | 18 | 24 | 29 | 21
  MTX: Medium dose (Baseline) (n=92,48,49,48,47) | 44 | 25 | 21 | 15 | 25
  MTX: High dose (Baseline) (n=92,48,49,48,47) | 9 | 5 | 4 | 4 | 1
  MTX: Increased (Day 1-85) (n=92,48,49,48,47) | 0 | 0 | 0 | 0 | 0
  MTX: No change (Day 1-85) (n=92,48,49,48,47) | 90 | 46 | 47 | 47 | 45
  MTX: Decreased (Day 1-85) (n=92,48,49,48,47) | 2 | 2 | 2 | 1 | 2
  MTX: Increased (Day 86-169) (n=85,45,46,48,45) | 2 | 3 | 3 | 2 | 1
  MTX: No change (Day 86-169) (n=85,45,46,48,45) | 82 | 42 | 42 | 46 | 44
  MTX: Decreased (Day 86-169) (n=85,45,46,48,45) | 1 | 0 | 1 | 0 | 0
  CST: Low dose (Baseline) (n=46,22,21,21,23) | 6 | 4 | 2 | 1 | 1
  CST: High dose (Baseline) (n=46,22,21,21,23) | 40 | 18 | 19 | 20 | 22
  CST: Increased (Day 1-85) (n=46,22,21,21,23) | 2 | 0 | 0 | 0 | 0
  CST: No change (Day 1-85) (n=46,22,21,21,23) | 44 | 22 | 21 | 21 | 23
  CST: Decreased (Day 1-85) (n=46,22,21,21,23) | 0 | 0 | 0 | 0 | 0
  CST: Increased (Day 86-169) (n=46,21,21,22,23) | 2 | 1 | 2 | 2 | 0
  CST: No change (Day 86-169) (n=46,21,21,22,23) | 44 | 20 | 19 | 20 | 23
  CST: Decreased (Day 86-169) (n=46,21,21,22,23) | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Mavrilimumab After First Dose by Region
Description: Data for European and Japanese regions were reported.
Time Frame: Blood samples were collected at pre-dose on Days 1, 4, 8, 15, 29, 57, and 85 as well as during follow up on Days 88, 99, 113 and 169
Population: The pharmacokinetic (PK) population included all participants who received mavrilimumab and for whom serum concentrations of mavrilimumab were available for PK data analyses. Here "N" signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for the specified region for each arm, respectively.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 46 | 49 | 49 | 45
nanogram per milliliter (ng/mL)
  European region (n=37,41,40,37) | 128 (1130) [43.0 to NA] | 917 (796) [29.0 to 58.0] | 1240 (1200) [42.0 to 89.0] | 6500 (3630) [29.0 to 45.0]
  Japanese region (n=9,8,9,8) | 61.3 (30.3) [NA to NA] | 633 (388) [NA to NA] | 1230 (652) [NA to NA] | 4540 (927) [NA to NA]

58. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for Mavrilimumab After First Dose by Region
Description: Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: The PK population included all participants who received mavrilimumab and for whom serum concentrations of mavrilimumab were available for PK data analyses. Here "N" signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for the specified region for each arm, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 46 | 49 | 49 | 45
days
  European region (n=37,41,40,37) | 4 (0.160) [2 to 7] | 3 (0.139) [2 to 12] | 4 (0.146) [0 to 8] | 4 (0.115) [2 to 8]
  Japanese region (n=9,8,9,8) | 6 (0.166) [2 to 8] | 7 (0.163) [3 to 9] | 6 (0.162) [2 to 9] | 7 (0.165) [2 to 8]

59. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Mavrilimumab After First Dose by Region
Description: Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: nanogram*day per milliliter (ng*day/mL)
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 46 | 49 | 49 | 45
nanogram*day per milliliter (ng*day/mL)
  European region (n=37,41,40,37) | 860 (8300) [43.0 to NA] | 6330 (5320) [29.0 to 58.0] | 10200 (10800) [42.0 to 89.0] | 62500 (36600) [29.0 to 45.0]
  Japanese region (n=9,8,9,8) | 504 (236) [NA to NA] | 5820 (4300) [NA to NA] | 11300 (6620) [NA to NA] | 45500 (12300) [NA to NA]

60. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Mavrilimumab After Last Dose by Region
Description: Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 42 | 40 | 45 | 45
ng/mL
  European region (n=33,33,37,37) | 137 (363) [43.0 to NA] | 1030 (3150) [29.0 to 58.0] | 2950 (2380) [42.0 to 89.0] | 7880 (5610) [29.0 to 45.0]
  Japanese region (n=9,7,8,8) | 136 (156) [NA to NA] | 1200 (727) [NA to NA] | 3340 (1290) [NA to NA] | 10300 (2470) [NA to NA]

61. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for Mavrilimumab After Last Dose by Region
Description: Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: as for outcome 58
Measure: Median (Full Range); unit: days
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 42 | 40 | 45 | 45
days
  European region (n=33,33,37,37) | 3 (0.160) [0 to 6] | 3 (0.139) [0 to 14] | 3 (0.146) [0 to 21] | 3 (0.115) [0 to 14]
  Japanese region (n=9,7,8,8) | 3 (0.166) [1 to 5] | 3 (0.163) [1 to 4] | 3.5 (0.162) [0 to 14] | 2 (0.165) [0 to 3]

62. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Mavrilimumab After Last Dose by Region
Description: Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 42 | 40 | 45 | 45
ng*day/mL
  European region (n=33,33,37,37) | 1060 (2770) [43.0 to NA] | 9260 (26300) [29.0 to 58.0] | 27900 (26700) [42.0 to 89.0] | 80500 (64300) [29.0 to 45.0]
  Japanese region (n=9,7,8,8) | 915 (1020) [NA to NA] | 12100 (9150) [NA to NA] | 34900 (18000) [NA to NA] | 104000 (30300) [NA to NA]

63. Secondary Outcome: Terminal Phase Elimination Half-Life (t1/2) for Mavrilimumab After Last Dose by Region
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 42 | 40 | 45 | 45
days
  European region (n=33,33,37,37) | 5.56 (4.08) [43.0 to NA] | 4.37 (2.88) [29.0 to 58.0] | 6.33 (3.07) [42.0 to 89.0] | 6.84 (3.00) [29.0 to 45.0]
  Japanese region (n=9,7,8,8) | 6.96 (4.61) [NA to NA] | 7.23 (5.67) [NA to NA] | 7.38 (1.65) [NA to NA] | 7.08 (2.19) [NA to NA]

64. Secondary Outcome: Accumulation Ratio for Mavrilimumab After Last Dose by Region
Description: Accumulation ratio was calculated as ratio of AUCtau after last dose and AUCtau after first dose. Data for European and Japanese regions were reported.
Time Frame: as for outcome 57
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 42 | 40 | 45 | 45
ratio
  European region (n=33,33,37,37) | 1.22 (2.97) [43.0 to NA] | 1.36 (2.23) [29.0 to 58.0] | 2.57 (54.1) [42.0 to 89.0] | 1.29 (0.932) [29.0 to 45.0]
  Japanese region (n=9,7,8,8) | 1.82 (1.85) [NA to NA] | 1.66 (0.716) [NA to NA] | 3.21 (3.21) [NA to NA] | 2.28 (0.616) [NA to NA]

65. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies (ADAs) to Mavrilimumab at Any Visit
Description: ADA detection measured by using electrochemiluminescence assays.
Time Frame: Day 1 up to Day 169
Population: The immunogenicity population included all participants who received at least 1 dose of CAM-3001 and for whom at least one serum sample for immunogenicity testing was available.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 10 mg | Mavrilimumab 30 mg | Mavrilimumab 50 mg | Mavrilimumab 100 mg
Number analyzed (Participants) | 96 | 48 | 49 | 49 | 48
participants | 3 (0.110) [57.0 to 88.0] | 10 (0.160) [43.0 to NA] | 6 (0.139) [29.0 to 58.0] | 2 (0.146) [42.0 to 89.0] | 2 (0.115) [29.0 to 45.0]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 169 (follow-up)
Groups:
- CAM-3001 10 MG: Mavrilimumab (CAM-3001) 10 milligram (mg) injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
- CAM-3001 30 MG: Mavrilimumab (CAM-3001) 30 mg injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
- CAM-3001 50 MG: Mavrilimumab (CAM-3001) 50 mg injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
- CAM-3001 100 MG: Mavrilimumab (CAM-3001) 100 mg injection subcutaneously every other week for 12 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) orally or parenterally.
Arm/Group | CAM-3001 10 MG | CAM-3001 30 MG | CAM-3001 50 MG | CAM-3001 100 MG | PLACEBO
Serious Adverse Events (participants affected / at risk) | 2/48 | 2/49 | 1/49 | 0/48 | 1/96
Other Adverse Events (participants affected / at risk) | 32/48 | 29/49 | 26/49 | 28/48 | 46/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM-3001 10 MG (N=48) | CAM-3001 30 MG (N=49) | CAM-3001 50 MG (N=49) | CAM-3001 100 MG (N=48) | PLACEBO (N=96)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM-3001 10 MG (N=48) | CAM-3001 30 MG (N=49) | CAM-3001 50 MG (N=49) | CAM-3001 100 MG (N=48) | PLACEBO (N=96)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth malformation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Injection site papule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infected bites (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (7) | 3 (3) | 5 (5) | 5 (5)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 4 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 10 (13) | 3 (3) | 5 (5) | 5 (6) | 5 (6)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nitrite urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spirometry abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 3 (4) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (5) | 0 (0) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Family stress (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Venous insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.